CLINICAL TRIAL: NCT02084836
Title: Relation of Consummatory & Anticipatory Food Reward to Obesity
Status: Completed | Type: Observational
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK080760; R01DK080760 (NIH)
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Obesity
Keywords: fMRI obesity adolescents
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lean adolescents
  Interventions: Other: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging

SUMMARY:
Obesity is associated with increased risk for mortality, atherosclerotic cerebrovascular disease, coronary heart disease, colorectal cancer, hyperlipidemia, hypertension, gallbladder disease, and diabetes mellitus, resulting in over 111,000 deaths annually in the United States (Calle et al., 1999; Flegal et al., 2005). In the US, 65% of adults are overweight or obese (Hedley et al., 2004). Unfortunately, the treatment of choice for obesity (behavioral weight loss treatment) only results in a 10% reduction in body weight on average and most patients regain this weight within a few years (Jeffery et al., 2000). Further, most obesity prevention programs do not reduce risk for future weight gain (Stice, Shaw, & Marti, 2006). The limited success of treatment and prevention interventions may be due to an incomplete understanding of the processes that increase risk for obesity. Recent data suggest that obese adults show abnormalities in reward from food intake and anticipated food intake relative to lean adults, but the precise nature of these abnormalities is unclear and it has not been established whether these abnormalities predate obesity onset or are a consequence. It is vital to elucidate risk factors for obesity onset to advance understanding of etiological processes and determine the content of prevention and treatment programs.

The goals of this study are to (1) determine whether adolescents at high-risk for obesity, by virtue of having two obese parents, show abnormalities in reward from food intake (consummatory food reward) and anticipated reward from food intake (anticipatory food reward) compared to adolescents who are at low-risk for obesity, (2) determine whether abnormalities in consummatory and anticipatory food reward increase risk for weight gain and obesity onset, (3) examine moderators that may amplify the relations of consummatory and anticipatory food reward to unhealthy weight gain, and (4) examine changes in consummatory and anticipatory food reward in those participants who show obesity onset relative to those not showing obesity onset.

ELIGIBILITY:
Inclusion Criteria:

* Between 14-17 years old
* BMI between 25th and 75th percentile

Exclusion Criteria:

* Contraindicators of functional magnetic resonance imaging (fMRI): metal implants, braces, pregnancy
* Symptoms of major psychiatric disorders (substance use disorders, conduct disorder, attention deficit hyperactive disorder, major depression, bipolar disorder, panic disorder, agoraphobia, generalized anxiety disorder) binge eating
* Current use of pyschoactive drugs
* Serious medical conditions (diabetes, brain injury)
* Current smoking
* Relevant food allergies
* Current weight loss dieting

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 162 lean adolescents between 14-17 years old with BMIs between the 25th and 75th percentile at baseline
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2009-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
increases in BMI | 1, 2, and 3 years
  To determine whether abnormalities in consummatory and anticipatory food reward increase risk for weight gain and obesity onset.

SECONDARY OUTCOMES:
(anticipated) reward from food intake | baseline
  To determine whether adolescents at high-risk for obesity, by virtue of having two obese parents, show abnormalities in reward from food intake (consummatory food reward) and anticipated reward from food intake (anticipatory food reward) compared to adolescents who are at low-risk for obesity.

OTHER OUTCOMES:
Changes in neural response to (anticipated) reward from food intake | baseline, 2, and 3 year
  Examine changes in consummatory and anticipatory food reward in those participants who show obesity onset relative to those not showing obesity onset

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Result] Stice E, Yokum S. Brain reward region responsivity of adolescents with and without parental substance use disorders. Psychol Addict Behav. 2014 Sep;28(3):805-15. doi: 10.1037/a0034460. Epub 2013 Oct 14. PMID 24128289
- [Result] Burger KS, Stice E. Elevated energy intake is correlated with hyperresponsivity in attentional, gustatory, and reward brain regions while anticipating palatable food receipt. Am J Clin Nutr. 2013 Jun;97(6):1188-94. doi: 10.3945/ajcn.112.055285. Epub 2013 Apr 17. PMID 23595877
- [Result] Stice E, Yokum S, Burger KS. Elevated reward region responsivity predicts future substance use onset but not overweight/obesity onset. Biol Psychiatry. 2013 May 1;73(9):869-76. doi: 10.1016/j.biopsych.2012.11.019. Epub 2013 Jan 8. PMID 23312561
- [Result] Stice E, Burger K, Yokum S. Caloric deprivation increases responsivity of attention and reward brain regions to intake, anticipated intake, and images of palatable foods. Neuroimage. 2013 Feb 15;67:322-30. doi: 10.1016/j.neuroimage.2012.11.028. Epub 2012 Nov 28. PMID 23201365
- [Result] Stice E, Yokum S, Burger K, Epstein L, Smolen A. Multilocus genetic composite reflecting dopamine signaling capacity predicts reward circuitry responsivity. J Neurosci. 2012 Jul 18;32(29):10093-100. doi: 10.1523/JNEUROSCI.1506-12.2012. PMID 22815523
- [Result] Burger KS, Stice E. Frequent ice cream consumption is associated with reduced striatal response to receipt of an ice cream-based milkshake. Am J Clin Nutr. 2012 Apr;95(4):810-7. doi: 10.3945/ajcn.111.027003. Epub 2012 Feb 15. PMID 22338036
- [Result] Stice E, Yokum S, Burger KS, Epstein LH, Small DM. Youth at risk for obesity show greater activation of striatal and somatosensory regions to food. J Neurosci. 2011 Mar 23;31(12):4360-6. doi: 10.1523/JNEUROSCI.6604-10.2011. PMID 21430137
- [Derived] Yokum S, Bohon C, Berkman E, Stice E. Test-retest reliability of functional MRI food receipt, anticipated receipt, and picture tasks. Am J Clin Nutr. 2021 Aug 2;114(2):764-779. doi: 10.1093/ajcn/nqab096. PMID 33851199
- [Derived] Hume DJ, Yokum S, Stice E. Low energy intake plus low energy expenditure (low energy flux), not energy surfeit, predicts future body fat gain. Am J Clin Nutr. 2016 Jun;103(6):1389-96. doi: 10.3945/ajcn.115.127753. Epub 2016 May 11. PMID 27169833
- [Derived] Stice E, Palmrose CA, Burger KS. Elevated BMI and Male Sex Are Associated with Greater Underreporting of Caloric Intake as Assessed by Doubly Labeled Water. J Nutr. 2015 Oct;145(10):2412-8. doi: 10.3945/jn.115.216366. Epub 2015 Sep 2. PMID 26338886
- [Derived] Stice E, Durant S. Elevated objectively measured but not self-reported energy intake predicts future weight gain in adolescents. Appetite. 2014 Oct;81:84-8. doi: 10.1016/j.appet.2014.06.012. Epub 2014 Jun 12. PMID 24930597